CLINICAL TRIAL: NCT00925249
Title: Comparison of the Tuberculin Skin Test (TST) and QuantiFERON ®-TB Gold Test (QFT-G) In Patients With Rheumatoid Arthritis Being Considered for Anti-TNF-Alpha Therapy
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Walter Reed Army Medical Center (U.S. Federal Agency)
Collaborators: National Naval Medical Center (U.S. Federal Agency)
Responsible Party: LT Robert O. Holmes JR D.O., US Navy Medical Corp
Other Study IDs: 6950
Record Dates: First submitted 2009-05-13; First posted 2009-06-22 (Estimated); Last update posted 2009-12-14 (Estimated); Status verified 2009-06

CONDITIONS: Rheumatoid Arthritis; Tuberculosis
Keywords: rheumatoid arthritis; RA; TB; tuberculosis; anti-TNF therapy; biologic therapy; quantiferon; IGRA; Newly diagnosed rheumatoid arthritis (RA) in the Tricare system
MeSH Terms: conditions — Arthritis, Rheumatoid; Tuberculosis

STUDY DESIGN:
Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- 1: The study group will consist of RA patients of the Walter Reed Army Medical Center (WRAMC) rheumatology clinic being considered for treatment with anti-TNF alpha therapy. We will enter patients into the study over a projected course of 12-24 months or until we reach the statistical requirement of 60 subjects.
- 2: The control group will consist of healthy subjects without known immune-dysregulation or history of treatment with biologic agents who present to the WRAMC Allergy- Immunology clinic for routine screening TST as a part of current WRAMC policy.

SUMMARY:
This research will help doctors interested in the usefulness of a new test to discover hidden tuberculosis infections in patients diagnosed with rheumatoid arthritis (RA). This new test is called Quantiferon-Gold (QFT-G). After immune system medicines that block TNF-alpha (a protein manufactured by white blood cells to stimulate and activate the immune system in response to infection or cancer) started to be used, the rate of tuberculosis infections in patients treated with these medicines has increased. Doctors think that the investigators may be missing some tuberculosis infections that were hidden before the medicine is started. This new QFT-G test might better diagnose these hidden tuberculosis infections than the current tuberculosis skin test, also known as a PPD/TST. The investigators would like to compare these two tests to find out which is better at detecting these hidden infections. At the same time the investigators will measure the strength of the patient's immune system with a blood test. If you are being considered for a TNF-alpha inhibitor medicine, or are getting the patient's routine PPD/TST, the investigators are asking for the patient's participation.

DETAILED DESCRIPTION:
In recent years the use of biologic agents for the treatment of rheumatic conditions has called into question the utility of the classic tuberculin skin test (TST) for the diagnosis of latent tuberculosis infection (LTBI). Current clinical rheumatology practice requires potential candidates of biologic therapy to have a negative TST before beginning biologic therapy. But since the TST is time consuming, operator dependent, and fraught with error, it may fail to alert physicians of LTBI in patients with autoimmune diseases and or pharmaceutical immunosuppression. Reactions to intradermal antigen placement requires many cellular interactions, but chiefly they must possess , a sufficient number of memory T cells, the ability to proliferate a clone of T cells specific to the antigen that is introduced, and the ability to traffic these effector cells to the local site. If any of these components are missing the individual may be unable to mount a type IV hypersensitivity (DTH-IV) reaction which is the basis for the TST. While many have recently compared the performance of the new IFN-gamma release assays (IGRAs) like the QuantiFERON-γ TB GOLD® (QFT-G) to the TST for the diagnosis of LTBI, no one has investigated the immunologic factors that may affect these results. Some have postulated that the QFT-G may be less affected by immune-suppression than the TST in patients with rheumatoid arthritis (RA). But recently this was called into question when significant numbers of indeterminate QFT-G results were seen in RA patients. Therefore, we plan to address two current clinical questions. First, what is the best screening strategy for LTBI in RA patients being started on biologic agents - TST, QFT-G or both? Second, is there utility in conducting immune competence testing in RA patients to predict those whom may be unable to generate a positive TST and/or QFT-G. This observational and exploratory pilot study will compare normal matched controls to RA patients being considered for anti-TNF alpha therapy. We will perform a comprehensive evaluation of the immune system by measuring memory T cell numbers with flow cytometry, the ability of memory T cells to proliferate to the tuberculin antigen or purified protein derivative (PPD), and phytohemagglutinin (PHA) antigen via the lymphocyte proliferation assay QunatiFERON-CMI.™ We will also investigate memory T cell trafficking ability via intradermal PPD and PHA antigen placement. Results of QFT-G tests will be compared to the TST with an emphasis on those results which are discordant. We will further attempt to identify immunocompetence testing which may help identify those patients who are unable to mount a DTH-IV response. In order to detect a statistical difference in this specific test population we will use analysis of variance for continuous or ordinal variables and the chi-square test (or Fisher exact test) for categorical data statistics. We hope to contribute to the body of literature regarding the best screening strategy for LTBI in patients with RA, and explore the concept of screening for immune competence in this specific population, which has not been elucidated in the literature.

ELIGIBILITY:
Inclusion Criteria:

Study group:

* Any patient 18 years or older who has been diagnosed with RA (American College of Rheumatology (ACR) criteria) and is being considered for de novo anti-TNF alpha therapy will be invited to participate in this study.

Control group:

* Control subjects will be any patient 18 years or older presenting to the Allergy/Immunology clinic for routine TST.

Exclusion Criteria:

Study group:

* We will exclude any individual with a previous history of known immuno-compromising disease state or unstable medical condition other than RA resulting in overall poor health and/or protein calorie deprivation to include:

  * any other autoimmune disease
  * oral steroid use in the past 3 days (4 half-lives of prednisone is 14 hours)
  * inhaled steroid use at a dose of > 2000 mg beclomethasone equivalent/day
  * any cancer [solid organ or blood]
  * radiation therapy in prior three months
  * any bleeding disorders
  * chemotherapeutic agents
  * transfusion or blood products in past 1 year
  * history of HIV
  * chronic hepatitis
  * malignancy
  * transplant history
  * chronic infection
  * chronic renal failure
  * current allergy treatment (shots, antihistamines)
  * uncontrolled diabetes, or the inability to provide informed consent
  * we will also exclude individuals with immediate hypersensitivity to the TST/PPD or PHA antigens
  * a previous severe local ulceration with TST/PPD
  * suspected active TB, previous TB treatment

Control group:

* We will exclude any individual with known history of anti-TNF alpha therapy.
* We will also exclude any patient with a history of any immune-modulatory (DMARD) therapy (steroids, anti-TNF agents, methotrexate, azathioprine, sulfasalazine, etc.) within the previous 12 months.
* Additionally we will exclude all those individuals with previous history of TB or TB therapy, diabetes mellitus, HIV, malignancy, or hepatitis that may influence the dermal reaction to PHA antigen or ex vivo CMI activity.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: patients in the US government tricare health system
Sampling Method: Probability Sample
Enrollment: 90 (Estimated)
Dates: Start 2009-05; Primary Completion 2011-05 (Estimated); Study Completion 2011-06 (Estimated)

PRIMARY OUTCOMES:
Primary endpoints are the results of the QFT-G test (defined as positive, negative or indeterminate) and the results of the TST (defined as positive or negative). | Patients will be enrolled over a 2 year time frame

SECONDARY OUTCOMES:
Secondary endpoints include the percentage and numbers of CD45RO (memory T cells), the response PHA intradermal antigen placement, numbers of hypoergic TSTs, and the results of cell mediated immunity (CMI) assays. | Patients will be enrolled over a 2 year time period

CONTACTS AND LOCATIONS:
Overall Officials: Adam T Armstrong, DO, Principal Investigator — Rheumatology Fellow - Walter Reed Army Medical Center; Robert O Holmes, DO, Study Chair — National Naval Medical Center
Locations (1):
- Walter Reed Army Medical Center, Washington D.C., District of Columbia, United States

REFERENCES:
- [Background] Greenberg JD, Reddy SM, Schloss SG, Kurucz OS, Bartlett SJ, Abramson SB, Bingham CO 3rd. Comparison of an in vitro tuberculosis interferon-gamma assay with delayed-type hypersensitivity testing for detection of latent Mycobacterium tuberculosis: a pilot study in rheumatoid arthritis. J Rheumatol. 2008 May;35(5):770-5. PMID 18322990
- [Background] Gomez-Reino JJ, Carmona L, Valverde VR, Mola EM, Montero MD; BIOBADASER Group. Treatment of rheumatoid arthritis with tumor necrosis factor inhibitors may predispose to significant increase in tuberculosis risk: a multicenter active-surveillance report. Arthritis Rheum. 2003 Aug;48(8):2122-7. doi: 10.1002/art.11137. PMID 12905464
- [Background] Carmona L, Gomez-Reino JJ, Rodriguez-Valverde V, Montero D, Pascual-Gomez E, Mola EM, Carreno L, Figueroa M; BIOBADASER Group. Effectiveness of recommendations to prevent reactivation of latent tuberculosis infection in patients treated with tumor necrosis factor antagonists. Arthritis Rheum. 2005 Jun;52(6):1766-72. doi: 10.1002/art.21043. PMID 15934089
- [Background] British Thoracic Society Standards of Care Committee. BTS recommendations for assessing risk and for managing Mycobacterium tuberculosis infection and disease in patients due to start anti-TNF-alpha treatment. Thorax. 2005 Oct;60(10):800-5. doi: 10.1136/thx.2005.046797. Epub 2005 Jul 29. PMID 16055611
- [Background] Matulis G, Juni P, Villiger PM, Gadola SD. Detection of latent tuberculosis in immunosuppressed patients with autoimmune diseases: performance of a Mycobacterium tuberculosis antigen-specific interferon gamma assay. Ann Rheum Dis. 2008 Jan;67(1):84-90. doi: 10.1136/ard.2007.070789. Epub 2007 Jul 20. PMID 17644549
- [Background] Takahashi H, Shigehara K, Yamamoto M, Suzuki C, Naishiro Y, Tamura Y, Hirohashi Y, Satoh N, Shijubo N, Shinomura Y, Imai K. Interferon gamma assay for detecting latent tuberculosis infection in rheumatoid arthritis patients during infliximab administration. Rheumatol Int. 2007 Oct;27(12):1143-8. doi: 10.1007/s00296-007-0361-2. Epub 2007 May 15. PMID 17503048
- [Background] Ponce de Leon D, Acevedo-Vasquez E, Sanchez-Torres A, Cucho M, Alfaro J, Perich R, Pastor C, Harrison J, Sanchez-Schwartz C. Attenuated response to purified protein derivative in patients with rheumatoid arthritis: study in a population with a high prevalence of tuberculosis. Ann Rheum Dis. 2005 Sep;64(9):1360-1. doi: 10.1136/ard.2004.029041. PMID 16100342
- [Background] D. Mines, Y. Gu, Q. Liu, L.N. Horne, M.J. Harrison. Global Safety Surveillance and Epidemiology. Wyeth Research, Collegeville, United States. [2008][OP-0138] Risk of Active Tuberculosis (TB) Among Biologic-Naïve RA Patients Retrospective Cohor Study in a US Claims Database. Ann Rheum Dis 2008;67(Suppl II):91.
- [Background] Chen DY, Shen GH, Hsieh TY, Hsieh CW, Lan JL. Effectiveness of the combination of a whole-blood interferon-gamma assay and the tuberculin skin test in detecting latent tuberculosis infection in rheumatoid arthritis patients receiving adalimumab therapy. Arthritis Rheum. 2008 Jun 15;59(6):800-6. doi: 10.1002/art.23705. PMID 18512714